CLINICAL TRIAL: NCT07199686
Title: Color Analysis of Graft and Recipient Site After Free Gingival Graft Surgery Using Polarized Digital Photograph
Brief Title: Digital Color Analysis of the Graft and Recipient Site After Free Gingival Graft Surgery
Status: Completed | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Other Study IDs: SKOLE; 2025\46 (Other: Bezmialem Vakif University Ethics Committee)
Record Dates: First submitted 2025-09-10; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Digital Photography; Cross Polarized Filter; Free Gingival Graft
Keywords: CIELab; Digital color analysis; cross-polarized filter; free gingival graft; gingiva color

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Clinical Periodontal Measurements and Digital Imaging: For each tooth within the FGG treated sites, probing pocket depth (PD), clinical attachment level (CAL), and keratinized gingiva width (KGW) were recorded. The thickness of the FGG and adjacent keratinized gingiva (KG) was assessed using a transgingival method. Standardized intraoral photographs were obtained from the study population.

SUMMARY:
This study evaluates gingival color following Free Gingival Graft (FGG) surgery using polarized digital photography to objectively analyze grafted and adjacent tissues. Conventional verbal descriptors (e.g., pale pink, salmon pink) lack precision; therefore, digital colorimetry provides objective, non-contact, and reproducible measurements. The protocol utilizes the CIELab system with standardized color disks and polarization to document postoperative color changes accurately.

The study objectives are: (1) to determine CIELab color values of FGG-treated gingiva in patients who underwent conventional surgery at least six months earlier; (2) to assess the influence of age, sex, time since surgery, and gingival thickness on these values; and (3) to compare graft color with adjacent gingiva.

Hypothesis: In FGG-treated patients, graft CIELab color values are unaffected by age, sex, postoperative duration, or gingival thickness.

DETAILED DESCRIPTION:
The aim of this cross-sectional study was to evaluate the color characteristics of free gingival graft (FGG) and the adjacent gingiva using polarized filtered digital photographs in cases where more than six months have elapsed since the procedure, and to assess the potential influence of clinical and sociodemographic factors on gingival color.

Fifty cases involving FGG procedures covering one or two lower anterior incisors were included in the study. Clinical parameters including probing pocket depth, bleeding on probing, clinical attachment level, width of keratinized gingiva, and thickness of keratinized gingiva were recorded. Standardized color reference disks were placed on the labial surfaces of the treated teeth, and both filtered and unfiltered photographs were taken. The images were saved in JPEG format and analyzed using the CIELab color system in Adobe Photoshop. A p-value of less than 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Postoperative period of at least 6 months after FGG
* Age between 18 and 65 years
* No known systemic diseases
* No use of medications adversely affecting gingival health (e.g., calcium channel blockers, immunosuppressants, antiepileptics)
* Full-mouth plaque index (PI)(1) and gingival index (GI)(2) < 1
* Probing pocket depth (PPD) ≤ 3 mm with no bleeding on probing (BOP)(3) in the mandibular anterior teeth
* Absence of habitual mouth breathing

Exclusion Criteria:

* Current smoking
* Pregnancy or lactation
* Previous endodontic or restorative treatment in the mandibular anterior teeth
* Parafunctional habits (e.g., bruxism) or history of orthodontic treatment
* Conditions impairing salivary flow (e.g., Sjögren's syndrome or similar disorders)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This retrospective cohort study included patients from the Department of Periodontology, Faculty of Dentistry, Bezmialem Vakıf University, who had undergone conventional free gingival graft (FGG) in the mandibular anterior region involving one or two teeth.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2023-03-20 (Actual); Primary Completion 2023-08-05 (Actual); Study Completion 2025-04-20 (Actual)

PRIMARY OUTCOMES:
Characterization of the color values of the Free Gingival Graft (FGG) according to the CIELab color system | Through study completion, an average of 6 months
  Standardized intraoral photographs were obtained from fifty participants. Digital images were obtained using a camera with standardized settings to ensure reproducibility. All images, taken with and without the filter. Photographs were analyzed in Adobe Photoshop programme using the CIELAB system. The FGG region was divided into three equal zones (coronal, middle, apical). For each region, mean L*, a*, and b* values were calculated.
Characterization of the color values of the adjacent keratinized gingiva according to the CIELab color system | Through study completion, an average of 6 months
  Standardized intraoral photographs were obtained from fifty participants. Digital images were obtained using a camera with standardized settings to ensure reproducibility. All images, taken with and without the filter. Photographs were analyzed in Adobe Photoshop programme using the CIELAB system. The adjacent keratized gingiva region was divided into two equal zones (coronal and middle) as the apical region corresponded to non-keratinized mucosa. For each region, mean L*, a*, and b* values were calculated.

SECONDARY OUTCOMES:
Keratinized Gingiva Width | Baseline
  For teeth within the operative area, the distance between the mucogingival junction and the gingival margin at the mesial, middle, and distal sites was measured. The mean of these three values was recorded as the keratinized gingiva width (KGW) for each tooth.
Periodontal pocket depth | Baseline
  Periodontal pocket depth (PPD) was measured as the distance from the gingival margin to the base of the pocket at the mesio-buccal, mid-buccal, and disto-buccal surfaces of each tooth in the operative region. The mean of these three measurements was recorded as the PPD value for the tooth.
Clinical attachment level | Baseline
  Clinical attachment level (CAL) was measured as the distance from the mesial, mid-buccal, and distal aspects of each tooth within the surgical area to the cemento-enamel junction (CEJ) and extended to the depth of the periodontal pocket. The mean of these three measurements was recorded, and the CAL for each tooth was determined accordingly.Time Frame:At the time of examination.
Measurement of gingival thickness | Baseline
  The thickness of the free gingival graft (FGG) and adjacent keratinized gingiva (KG) was assessed using a transgingival probing method. After administering local anesthesia, a #25 endodontic spreader was inserted perpendicularly through the mucosa until it contacted the underlying hard tissue. The distance between the spreader tip and the stopper was measured with a digital caliper. In the FGG area, measurements were obtained at three points (mesial, middle, and distal). In the adjacent keratinized tissue, two measurements were taken 2 mm apical to the gingival margin of the neighboring tooth, corresponding to the coronal and mid-regions of the graft.
Influence of age on color values | Through study completion, an average of 6 months
  Patient age was recorded, and the effect of age (year) on the CIELab values of the graft was assessed via One way Multivariate Analysis of Variance.
Influence of 'time since surgery' on color values | Through study completion, an average of 6 months
  The duration 'since FGG surgery (months)' was recorded, and its effect on the CIELab values of the graft was assessed via One way Multivariate Analysis of Variance.
Influence of gender on color values | Through study completion, an average of 6 months
  Patient gender (female/male) was recorded, and the effect of gender (female/male) on the CIELab values of the graft was assessed via One way Multivariate Analysis of Variance.
Influence of gingival thickness on color values | Through study completion, an average of 6 months
  Gingival thickness was recorded, and the effect of gingival thickness (mm) on the CIELab values of the graft was assessed via One way Multivariate Analysis of Variance

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakif University, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available upon publication of the manuscript